CLINICAL TRIAL: NCT05332288
Title: Triphasic Osteochondral Scaffold for the Treatment of Osteochondritis Dissecans of the Knee: Observational Study
Brief Title: Triphasic Osteochondral Scaffold for the Treatment of the OCD of the Knee: Observational Study
Acronym: MAIOCD
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: MAIOCD
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Osteochondritis Dissecans Knee
Keywords: knee; OCD; Osteochondritis dissecans; scaffold; Maioregen; biomimetic; Osteochondral lesions
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the present study is to evaluate the clinical results of reconstructive treatment of knee OCD defects treated with osteochondral scaffolds implanted with specific instrumentation.The evaluation will be performed through clinical, subjective and objective assessments.

DETAILED DESCRIPTION:
30 patients affected by OCD of the knee will be included in observational, perspective, monocentric trial. Patients will undergo clinical follow-up visits and administration of questionnaires before surgery and at 6, 12, 24 and 60 months after surgery. A CRF (Case Report Form) related to the patient's specific evaluation will be completed for each visit. Patients will also have imaging (MRI) examinations before surgery and at 12, 24 and 60 months after surgery as per normal clinical practice. Evaluation of the quality of cartilage repair will be assessed by specific MRI radiographic scores.

ELIGIBILITY:
Inclusion Criteria

* Male or female patients, aged 15-40 years;
* Single symptomatic osteochondral injury from OCD classified as ICRS OCD III or IV at the level of the femoral condyles;
* Failure of conservative treatment
* Lesion size between 1 and 10 cm2;
* BMI ≤ 30;
* Ability and consent of patients to actively participate in the rehabilitation protocol and clinical and radiological follow-up.

Exclusion Criteria:

* -Additional grade III or IV cartilage injury on the knee being treated;
* Advanced osteoarthritis
* Systemic or localized infection
* Systemic (e.g. rheumatoid arthritis) or local (e.g. synovitis) inflammatory diseases and cardiovascular diseases
* Immune system disorders
* Degenerative or vascular bone pathology (e.g. osteonecrosis)
* Coagulation disorders
* Systemic conditions that alter wound healing
* Established allergy to equine collagen and calcium phosphate salts
* Presence of ligamentous/patellofemoral instability/malignment, varus or valgus malalignment ≤ 3° that cannot be treated/corrected simultaneously;
* Previous tendon repair, ligamentous reconstruction, or realignment procedures within the past 12 months;
* Presence of any known human immunodeficiency virus, hepatitis, syphilis, malignant neoplasms and ongoing anti-neoplastic chemotherapy and radiation treatment; Uncontrolled diabetes; Uncontrolled thyroid function changes; Uncontrolled metabolic disorders; Renal disease and hypercalcemia
* Uncooperative patients, including those with a history of alcohol and drug abuse; Participation in another clinical trial or medical device trial that clinically interferes with the present pilot study;
* Incapacitated patients;
* Pregnant or lactating women. In particular, in the case of a suspected pregnancy in a patient of childbearing age, this will be excluded by serological testing (hCG).

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with knee OCD (ICRS OCD 3-4) with surgical indication for treatment of these lesions by biological reconstructive technique with osteochondral scaffolds will be enrolled. The estimated number of patients enrolled is 30, of which we expect from epidemiological data that about one third (10 patients) are between 15 and 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
IKDC-Subjective Score | 24 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function

SECONDARY OUTCOMES:
IKDC-Subjective Score | baseline, 6 months, 12 months, 60 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function
IKDC-Objective Score | baseline, 6 months, 12 months, 24 months, 60 months
  The objective rating scale has seven parameters related to knee function. The presence of effusions and degree of knee motion are assessed; the worst value of any of these parameters determines the final IKDC grade. There are four grades (A, B, C, D) that identify a knee rated as normal, near normal, abnormal, and severely abnormal, respectively;
KOOS Score | baseline, 6 months, 12 months, 24 months, 60 months
  KOOS SCORE consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items).
TegnerActivity Level Scale | baseline, 6 months, 12 months, 24 months, 60 months
  Tegner activity level scale allows to know the level of physical activity carried out by the patients. Tegner's activity scale classifies the activity according to work and sports activities on a scale from 0 to 10. Zero represents disability because of knee problems and 10 represents soccer a national or international level
EQ-5D (EuroQoL) Current Health Assessment | baseline, 6 months, 12 months, 24 months, 60 months
  The EQ-5D profile, asks patients to classify their health based on self-assessed levels of problems ("no", "some", "extreme") on five dimensions.
Patient Acceptable Symptom State (PASS | baseline, 6 months, 12 months, 24 months, 60 months
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no"
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score | 12 months, 24 months, 60 months
  The MOCART score 2.0 is a data point of interest because it allows for the assessment of both the repair of the specific cartilage tissue and the structures surrounding it. The MOCART score 2.0 is based on nine variables measured on a standard MRI and summed to a score, ranging from 0 to 100, where 100 represents the best score and a score of 0 represents the worst score. The underlying factors that may influence the MOCART 2.0 score are the severity of the defect prior to cartilage repair surgery;

CONTACTS AND LOCATIONS:
Overall Officials: Luca Andriolo, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriolo L, Crawford DC, Reale D, Zaffagnini S, Candrian C, Cavicchioli A, Filardo G. Osteochondritis Dissecans of the Knee: Etiology and Pathogenetic Mechanisms. A Systematic Review. Cartilage. 2020 Jul;11(3):273-290. doi: 10.1177/1947603518786557. Epub 2018 Jul 12. PMID 29998741
- [Background] Andriolo L, Candrian C, Papio T, Cavicchioli A, Perdisa F, Filardo G. Osteochondritis Dissecans of the Knee - Conservative Treatment Strategies: A Systematic Review. Cartilage. 2019 Jul;10(3):267-277. doi: 10.1177/1947603518758435. Epub 2018 Feb 22. PMID 29468901
- [Background] Filardo G, Andriolo L, Soler F, Berruto M, Ferrua P, Verdonk P, Rongieras F, Crawford DC. Treatment of unstable knee osteochondritis dissecans in the young adult: results and limitations of surgical strategies-The advantages of allografts to address an osteochondral challenge. Knee Surg Sports Traumatol Arthrosc. 2019 Jun;27(6):1726-1738. doi: 10.1007/s00167-018-5316-5. Epub 2018 Dec 6. PMID 30523367
- [Background] Andriolo L, Di Martino A, Altamura SA, Boffa A, Poggi A, Busacca M, Zaffagnini S, Filardo G. Matrix-assisted chondrocyte transplantation with bone grafting for knee osteochondritis dissecans: stable results at 12 years. Knee Surg Sports Traumatol Arthrosc. 2021 Jun;29(6):1830-1840. doi: 10.1007/s00167-020-06230-y. Epub 2020 Aug 18. PMID 32809120
- [Background] Minas T, Ogura T, Headrick J, Bryant T. Autologous Chondrocyte Implantation "Sandwich" Technique Compared With Autologous Bone Grafting for Deep Osteochondral Lesions in the Knee. Am J Sports Med. 2018 Feb;46(2):322-332. doi: 10.1177/0363546517738000. Epub 2017 Nov 10. PMID 29125919
- [Background] Boffa A, Solaro L, Poggi A, Andriolo L, Reale D, Di Martino A. Multi-layer cell-free scaffolds for osteochondral defects of the knee: a systematic review and meta-analysis of clinical evidence. J Exp Orthop. 2021 Jul 30;8(1):56. doi: 10.1186/s40634-021-00377-4. PMID 34331140
- [Background] Kon E, Filardo G, Brittberg M, Busacca M, Condello V, Engebretsen L, Marlovits S, Niemeyer P, Platzer P, Posthumus M, Verdonk P, Verdonk R, Victor J, van der Merwe W, Widuchowski W, Zorzi C, Marcacci M. A multilayer biomaterial for osteochondral regeneration shows superiority vs microfractures for the treatment of osteochondral lesions in a multicentre randomized trial at 2 years. Knee Surg Sports Traumatol Arthrosc. 2018 Sep;26(9):2704-2715. doi: 10.1007/s00167-017-4707-3. Epub 2017 Sep 14. PMID 28913600
- [Background] Di Martino A, Perdisa F, Filardo G, Busacca M, Kon E, Marcacci M, Zaffagnini S. Cell-Free Biomimetic Osteochondral Scaffold for the Treatment of Knee Lesions: Clinical and Imaging Results at 10-Year Follow-up. Am J Sports Med. 2021 Aug;49(10):2645-2650. doi: 10.1177/03635465211029292. Epub 2021 Jul 20. PMID 34283948
- [Background] Sessa A, Perdisa F, Di Martino A, Zaffagnini S, Filardo G. Cell-Free Biomimetic Osteochondral Scaffold: Implantation Technique. JBJS Essent Surg Tech. 2019 Aug 14;9(3):e27. doi: 10.2106/JBJS.ST.18.00089. eCollection 2019 Jul-Sep. PMID 32021725